CLINICAL TRIAL: NCT06237348
Title: Airway Clearance Therapy With Simeox Technology in Non-Cystic Fibrosis Bronchiectasis Patients With Chronic Mucus Hypersecretion - A Multicenter Randomized Controlled Trial Pilot Study
Brief Title: Simeox Therapy at Home Versus Standard of Care in NCFB Patients With CMH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Physio-Assist (Industry)
Collaborators: Medical University of Lodz (Other); University Hospital in Krakow (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Simeox 1.1 290623
Record Dates: First submitted 2024-01-11; First posted 2024-02-01 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Non-cystic Fibrosis Bronchiectasis; Chronic Mucus Hypersecretion
Keywords: NCFB; CMH; Simeox; Airway clearance; ACT; Bronchiectasis; Telecare
MeSH Terms: conditions — Bronchiectasis | interventions — Breathing Exercises

STUDY DESIGN:
Intervention Model Description: Prospective, open-label, parallel, Multicenter Randomized controlled trial,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Simeox (Experimental): Airway clearance device
  Interventions: Device: Simeox; Combination Product: Control
- Control (Active Comparator): Usual chest physiotherapy (manual, breathing exercise, PEP/oPEP)
  Interventions: Combination Product: Control

INTERVENTIONS:
Device: Simeox — Daily airway clearance therapy at home during 2 months
  Arms: Simeox
Combination Product: Control — Daily airway clearance therapy at home during 2 months
  Other Names: Usual chest physiotherapy (manual, breathing exercise, PEP/oPEP)

SUMMARY:
This pilot RCT will assess benefits of Simeox technology on lung function, respiratory symptoms, health-related quality of life, subjective efficiency, device adherence at home, Patient satisfaction, tolerance, safety, and telecare feasibility.

DETAILED DESCRIPTION:
Non-cystic fibrosis bronchiectasis (NCFB) is a chronic respiratory disease with multiple etiologies characterized by an irreversible dilatation of bronchi and an impair mucociliary clearance. These alterations cause sticky mucus retention and leads to recurrent infections and chronic bronchial inflammations. Chest physiotherapy is one of the cornerstones of the management of NCFB patients, particularly to facilitate airway clearance. In NCFB patients with chronic mucus hypersecretion (CMH), it is recommended that airway clearance sessions be carried out daily or several times a day, which represents a very significant burden of care. Moreover, access to respiratory physiotherapy for patients can be limited due to several causes: geographical, time or healthcare professional availability constraints. In addition, few healthcare professionals are trained for bronchial drainage especially with airway clearance devices.

SIMEOX® (Physio-Assist, France) is an innovative medical device (CE medical mark) for mucus clearance. The device is connected to patient mouth with an expiratory kit circuit. When the patient starts up the device during exhalation only, SIMEOX® disseminates a vibratory pneumatic signal in the bronchi that liquefies mucus and transports it from distal to central airways for sputum expectoration. After device training with respiratory physiotherapist, patients can be treated at hospital and use SIMEOX® in autonomy at home. Device training and patient follow-up can be performed also remotely with telecare with similar efficiency than face to face visits with health care professionals.

The main objective of this Pilot study is to evaluate the effects of mid-term use of SIMEOX® in autonomy at home for 2 months in NCFB patients with CMH and pulmonary exacerbation (in- or outpatients) in comparison to standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Patient with confirmed diagnosis of bronchiectasis confirmed by High Resolution Computed Tomography (HRCT): idiopathic, post-infective, systemic disease, ABPA, asthma, COPD, PCD
* Overproduction of mucus (ie: estimated bronchorrhea >10mL/day).
* Pulmonary exacerbation (in- or outpatients)
* Age > 18 years old
* Patient able to understand the study and to perform the 2-month follow up visit

Exclusion Criteria:

* Pneumothorax/pneumo-mediastinum in the six months prior hospitalization
* Recent episode of severe haemoptysis
* Unstable severe cardiac disease or hemodynamic instability
* Cystic fibrosis or COPD as dominant diagnosis
* Patient on lung transplant list
* Severe lung injuries
* Recent lung surgery
* Inhalation support (continuous ventilatory support)
* Tracheostomy
* Uncontrolled GERD
* Any contraindication to an instrumental bronchial clearance technique (up to the investigator)
* Inability to perform PFT or 6MWT
* Patient not available or wishing to move to a different region within 2 months of inclusion
* Patient considered by the investigator to be physically or mentally inapt to use the device and/or to perform the study procedures.
* Patient currently participating or having participated within one month prior to inclusion in a clinical intervention research trial that may impact the study, the impact of which is up to the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-10-15 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
To describe the evolution in Self-reported home adherence from baseline (hospital discharge) during follow-up | 2 months
  The evolution of device adherence will be described by % of self-reported sessions (0-1; 2-3; 4-7/week) by the patient over the 2-month FU (1 week, 2 weeks, 1 month and 2 months)

SECONDARY OUTCOMES:
To describe Simeox therapy settings (program selection) during follow-up | 2 months
  Simeox settings will be described by program selection (1, 2 or 3)
To describe Simeox therapy settings (intensity) during follow-up | 2 months
  Simeox settings will be described by intensity (25%, 50%, 75% or 100%)
To describe Simeox therapy settings (number of session) during follow-up | 2 months
  Simeox settings will be described by the number of sessions per day
To describe Simeox therapy settings (session duration) during follow-up | 2 months
  Simeox settings will be described by the session duration in minutes
To evaluate mucus quality with Simeox therapy during follow-up | 2 months
  Mucus quality will be evaluated during follow-up with a score from 1 to 4 (abondant - Scanty)
To evaluate breathing quality with Simeox therapy during follow-up | 2 months
  Breathing quality level will be evaluated during follow-up with a score from 1 to 4 (very good - very poor)
To evaluate ease handling of the Simeox device during follow-up | 2 months
  Ease of handling level will be evaluated during follow-up with a score 1 to 4 (very easy - not easy at all)
To evaluate pain during Simeox therapy | 2 months
  Pain level will be evaluated during follow-up with a scale from 0 to10 (no painful - very painful)
To evaluate fatigue during Simeox therapy | 2 months
  Fatigue level will be evaluated during follow-up with a scale from 0 to 10 (no fatigue - very tired)
To evaluate ease of use of Simeox device after 2 months of therapy | 2 months
  Ease of use level will be evaluated at 2 month with a score from 1 to 4 (very easy - not easy at all)
To evaluate patient preference between Simeox device and usual care after 2 months of therapy | 2 months
  Patient preference will be evaluated at 2 month in comparaison to conventional techniques used (yes/no)
To evaluate patient recommendation to others patients of Simeox device after 2 months of therapy | 2 months
  Patient recommendation to others patients will be evaluated at 2 month (yes/no)
Evaluate the feasibility of telecare during follow-up | 2 months
  Feasibility of telecare during follow-up will be estimated by the percent of call visit performed with the patients compared to the number of call visits scheduled in the protocol
To evaluate the effect of Simeox on respiratory symptoms in NCFB patients after 2 months of therapy | 2 months
  The change in respiratory symptoms score from baseline (hospital discharge) to 2-month FU will be measured with the Chronic Airways Assessment Test (CAT) questionaire
To evaluate the effect of Simeox on the health-related quality of life of NCFB patients after 2 months of therapy | 2 months
  The change in quality of life from baseline (hospital discharge) to 2-month FU will be measured with the St Georges Respiratory Questionnaire (SGRQ)
To evaluate the effect of Simeox on Forced Expiratory Volume at 1 seconde (FEV1) after 2 monts of therapy | 2 months
  The change in FEV1 from baseline (hospital discharge) to 2-month FU will be measured with spirometry
To evaluate the effect of Simeox on Forced Vital Capacity (FVC) after 2 monts of therapy | 2 months
  The change in FVC from baseline (hospital discharge) to 2-month FU will be measured with spirometry
To evaluate the effect of Simeox on Forced Expiratory Flow (FEF) at 25%, 50% and 75% of FVC after 2 monts of therapy | 2 months
  The change in FEF at 25%, 50% and 75% from baseline (hospital discharge) to 2-month FU will be measured with spirometry
To evaluate the effect of Simeox on dyspnea after 2 monts of therapy | 2 months
  The change in dyspnea from baseline (hospital discharge) to 2-month FU will be measured with the modified Medical Research Council (mMRC) questionnaire
To evaluate the effect of Simeox on exercise capacity after 2 monts of therapy | 2 months
  The change in walking distance from baseline (hospital discharge) to 2-month FU will be measured with the 6-min walking test (6MWT)
To evaluate safety of Simeox | 2 months
  The safety of Simeox will be assessed by the rate and severity of Side effects during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Wojciech PIOTROWSKI, MD, PhD, Study Director — Medical University of Lodz
Locations (2):
- Poland (2):
  - Jagiellonian University Medical College, Krakow
  - N. Barlicki University Hospital No 1, Lodz